CLINICAL TRIAL: NCT00322868
Title: A Pilot Study Assessing the Safety and Efficacy of Pioglitazone as an Anti-inflammatory Agent for the Treatment of CF Lung Disease in Patients With Cystic Fibrosis
Brief Title: Safety and Efficacy of Pioglitazone as an Anti-inflammatory for the Treatment of Cystic Fibrosis (CF) Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Michael W. Konstan, Professor of Pediatrics, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFFTI-Pio001
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Cystic Fibrosis
Keywords: Prescription drugs; Administration, oral; Durable medical equipment; Kinetics
MeSH Terms: conditions — Cystic Fibrosis | interventions — Pioglitazone

STUDY DESIGN:
Masking Description: This was open-label and no one was masked.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitazone (Experimental): All subjects treated for 28 days with pioglitazone, 30 mg orally, once daily Other names: Actos, Takeda
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: pioglitazone — All subjects treated for 28 days with pioglitazone, 30 mg orally, once daily.
  Other Names: Actos; Takeda

SUMMARY:
Study Hypothesis: Pioglitazone may decrease inflammation in cystic fibrosis lung disease.

Primary outcomes: Markers of inflammation (neutrophils, elastase, cytokines and bacteria)will be measured in induced sputum specimens before and after a 4 week treatment period with pioglitazone in clinically stable CF patients.

DETAILED DESCRIPTION:
* Single-center, open label study of pioglitazone in clinically stable patients with mild to moderate CF lung disease
* Induced sputum will be obtained from each subject at enrollment (Baseline) and again following 28 days of pioglitazone treatment (End of Treatment)
* Changes in markers of inflammation in the sputum samples will be assessed
* Safety measures, including complete blood count (CBC), serum chemistry, Erythrocyte sedimentation rate (ESR), C-Reactive Protein (CRP), urinalysis and spirometry, will also be assessed

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 28 years of age
* Confirmed diagnosis of cystic fibrosis
* Forced Expiratory Volume in 1 second (FEV1) >= 40% predicted
* Clinically stable
* Ability to reproduce spirometry
* Ability to understand and sign the informed consent

Exclusion Criteria:

* Use of an investigational agent within 4-week period prior to Visit 1
* Chronic daily use of ibuprofen or other NSAIDS
* Chronic daily use of insulin,oral diabetic agents or oral hypoglycemic agents
* History of hypersensitivity to beta agonists
* History of hypersensitivity to glitazones
* Oxygen saturation<92%
* Pregnant, breastfeeding or unwilling to practice acceptable birth control
* History of hemoptysis >30cc per episode within 30 days prior to Visit 1
* Significant history of hepatic, cardiovascular, renal,neurologic, hematologic or peptic ulcer disease
* Serum Glutamic-Oxaloacetic Transaminase (SGOT)/(Serum Glutamic Pyruvic Transaminase (SGPT) >3 times the upper limit of normal at screening, documented biliary cirrhosis,or portal hypertension
* Creatinine > 1.8 mg/dL at screening
* Inability to swallow pills
* Presence or abnormality that in the opinion of the investigator would compromise the safety or the quality of the data
* Subjects who have routinely taken ibuprofen or other NSAIDS; prednisone or other systemic corticosteroids, or insulin, or oral diabetic agents within 4 weeks prior to visit 1 or who have taken these medications as needed within 72 hours prior to visit one will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Konstan, MD, Principal Investigator — Case University and Rainbow Babies and Children's Hospital
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individualized personal data (IPD) will not be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients who will be approached for participation in this trial will first be identified using either Port CF (CFF Registry) or CF Center database. Once potentials are identified a chart review will be conducted to determine eligibility. Patients will approached at clinic for possible participation in the study.
Pre-assignment Details: Washout: A 4 week washout from chronic use of NSAIDs, corticosteroids and oral meds to treat diabetes will be required. Subjects will be excluded if they take these medication within 72 hours of Visit 1. Subjects using alternate month tobramycin for inhalation (TOBI) will need to be on an off cycle to participate in this study.
Groups:
- Pioglitazone (30 mg): After screening eligibility requirements were met, cystic fibrosis subjects received pioglitazone orally, 30 mg, once daily, for 28 days
Period: Overall Study
Arm/Group | Pioglitazone (30 mg)
Started | 21
Completed | 20
Not Completed | 1
Not completed — disease progression | 1

BASELINE CHARACTERISTICS:
Population: 21 subjects were screened and enrolled with 1 subject withdrawal due to disease progression.
Arm/Group | Pioglitazone (30 mg)
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — great or equal to 18 years of age Population: 1 subject withdrawn due to disease progression
  years
    number analyzed (Participants) | 20
    (all) | 30 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 subject was withdrawn and no samples analyzed
  Participants
    number analyzed (Participants) | 20
    Female | 8
    Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 subject withdrawn due to disease progression. no samples analyzed.
  Participants
    number analyzed (Participants) | 20
    Hispanic or Latino | 0
    Not Hispanic or Latino | 20
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 subject withdrawn due to disease progression no samples analyzed
  Participants
    number analyzed (Participants) | 20
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 18
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: 1 subject was withdrawn due to disease progression. No samples analyzed.
  Participants
    United States: number analyzed (Participants) | 20
    United States | 20
Total white cell count [Mean (Standard Deviation); unit: log 10 (cells/mL)] — Population: 1 subject withdrawn due to disease progression. No samples analyzed.
  log 10 (cells/mL)
    number analyzed (Participants) | 20
    (all) | 6.93 (0.40)
Total neutrophil count [Mean (Standard Deviation); unit: Log 10 (PMN/mL)] — Population: 1 subject withdrawn due to disease progression. No samples analyzed.
  Log 10 (PMN/mL)
    number analyzed (Participants) | 20
    (all) | 6.88 (0.39)
percent neutrophils [Mean (Standard Deviation); unit: percent of white blood cells] — Population: 1 subject withdrawn due to disease progression. No samples analyzed
  percent of white blood cells
    number analyzed (Participants) | 20
    (all) | 82.47 (11.88)

OUTCOME MEASURES:

1. Primary Outcome: Sputum White Cell Count
Description: The total number of white cells log 10 cells/mL
Time Frame: Day 0 and Day 29
Population: Of the 20 enrolled subjects, one did not produce sputum at Baseline and a second subject's Post-Treatment sputum sample was lost due to a lab error. This reduced the number of subjects per group to 19. Of these 19 subjects, 18 subjects had both Baseline and Post-Treatment sputum samples.
Measure: Mean (Standard Deviation); unit: log 10 (cells/mL)
Groups:
- Baseline: Results pre-Pioglitazone dosing
- Post-Treatment: Results following 28 days of Pioglitazone (oral, 30mg, once daily)
Arm/Group | Baseline | Post-Treatment
Number analyzed (Participants) | 19 | 19
log 10 (cells/mL) | 6.93 (0.40) | 6.81 (0.41)
Statistical Analysis 1: Comparison: Baseline vs Post-Treatment; Test type: Superiority or Other; p = 0.2772, t-test, 1 sided; Paired t-test analysis of the intra-subject change in log10 sputum white cell count

2. Primary Outcome: Sputum Neutrophil Count
Description: sputum neutrophils log 10 (cells/mL)
Time Frame: Day 0 and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log 10 (cells/mL)
Arm/Group | Baseline | Post-Treatment
Number analyzed (Participants) | 19 | 19
log 10 (cells/mL) | 6.88 (0.39) | 6.75 (0.42)
Statistical Analysis 1: Comparison: Baseline vs Post-Treatment; Test type: Superiority or Other; p = 0.2467, t-test, 1 sided; Paired t-test analysis of the intra-subject change in log10 sputum neutrophil count

3. Primary Outcome: Sputum Neutrophil Percent
Description: Neutrophils as a percent of the total white cells.
Time Frame: Day 0 and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent (%) of white blood cells
Arm/Group | Baseline | Post-Treatment
Number analyzed (Participants) | 19 | 19
Percent (%) of white blood cells | 82.47 (11.88) | 74.44 (17.07)
Statistical Analysis 1: Comparison: Baseline vs Post-Treatment; Test type: Superiority or Other; p = 0.0288, t-test, 1 sided; Paired t-test analysis of the intra-subject change in sputum percent neutrophils

4. Primary Outcome: Sputum Active Elastase
Description: Log 10 of Concentration of active Elastase in mcg/mL
Time Frame: Day 0 and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log 10 (mcg/mL)
Arm/Group | Baseline | Post-Treatment
Number analyzed (Participants) | 19 | 19
log 10 (mcg/mL) | 2.03 (0.36) | 1.96 (0.36)
Statistical Analysis 1: Comparison: Baseline vs Post-Treatment; Test type: Superiority or Other; p = 0.50, t-test, 1 sided; Paired t-test analysis of the intra-subject change in log10 sputum active elastase

5. Primary Outcome: Sputum TNFα
Description: The concentration of Tumor Necrosis Factor-α (TNFα) log 10 (pg/mL)
Time Frame: Day 0 and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log 10 (pg/mL)
Arm/Group | Baseline | Post-Treatment
Number analyzed (Participants) | 19 | 19
log 10 (pg/mL) | 1.74 (0.49) | 1.69 (0.59)
Statistical Analysis 1: Comparison: Baseline vs Post-Treatment; Test type: Superiority or Other; p = 0.62, t-test, 1 sided; Paired t-test analysis of the intra-subject change in log10 sputum TNFα

6. Primary Outcome: Sputum IL-1ß
Description: The concentration of Interleukin-1ß (IL-1ß) log 10 (pg/mL)
Time Frame: Day 0 and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log 10 (pg/mL)
Arm/Group | Baseline | Post-Treatment
Number analyzed (Participants) | 19 | 19
log 10 (pg/mL) | 4.05 (0.42) | 3.99 (0.52)
Statistical Analysis 1: Comparison: Baseline vs Post-Treatment; Test type: Superiority or Other; p = 0.50, t-test, 1 sided; Paired t-test analysis of the intra-subject change in log10 sputum IL-1ß

7. Primary Outcome: Sputum IL-6
Description: The concentration of Interleukin-6 (IL-6) log 10 (pg/mL)
Time Frame: Day 0 and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log 10 (pg/mL)
Arm/Group | Baseline | Post-Treatment
Number analyzed (Participants) | 19 | 19
log 10 (pg/mL) | 1.38 (0.33) | 1.41 (0.32)
Statistical Analysis 1: Comparison: Baseline vs Post-Treatment; Test type: Superiority or Other; p = 0.55, t-test, 1 sided; Paired t-test analysis of the intra-subject change in log10 sputum IL-6

8. Primary Outcome: Sputum IL-8
Description: Concentration of Interleukin-8 log 10 (pg/mL)
Time Frame: Day 0 and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log 10 (pg/mL)
Arm/Group | Baseline | Post-Treatment
Number analyzed (Participants) | 19 | 19
log 10 (pg/mL) | 5.13 (0.35) | 5.10 (0.34)
Statistical Analysis 1: Comparison: Baseline vs Post-Treatment; Test type: Superiority or Other; p = 0.75, t-test, 1 sided; Paired t-test analysis of the intra-subject change in log10 sputum IL-8

ADVERSE EVENTS:
Groups:
- Pioglitazone (30 mg): After screening eligibility requirements were met, cystic fibrosis subjects received pioglitazone orally,30 mg, once daily for 28 days
Arm/Group | Pioglitazone (30 mg)
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (30 mg) (N=20)
hypoglycemic event (Endocrine disorders) | 1 — Non serious, unexpected, possibly study related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No